CLINICAL TRIAL: NCT02257827
Title: Randomized Trial Comparing Intensity Modulated Radiotherapy Versus Conformal Radiotherapy to Treat Prostate Cancer With Hypofractionated Schedule.
Brief Title: Trial Comparing Intensity Modulated Radiotherapy Versus Conformal Radiotherapy to Treat Prostate Cancer With Hypofractionated Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustavo Viani Arruda (Other)
Responsible Party: Sponsor-Investigator, Gustavo Viani Arruda, Gustavo Arruda Viani, M.D, Phd., Marilia Medicine School
Organization: Marilia Medicine School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMEMA-0913
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
Keywords: Hypofractionated schedule; Intensity Modulated Radiotherapy; Conformal radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMRT- Hypofractionated schedule 70 Gy/25 fx (Experimental): The IMRT plan consisted of five - seven fields to deliver the same dose prescribed at the isodose line covering 95% of PTV.By the linear-quadratic formula, considering an α/β ratio of 1.5 Gy for prostate cancer, 70 Gy/25 fractions is equivalent to 86 Gy in 43 fractions of 2 Gy. All patients were simulated on CT simulator.
  Interventions: Radiation: IMRT
- 3DCRT-Hypofractionated schedule 70 Gy/25 fx (Active Comparator): The 3DCRT plan consisted of six fields to deliver a total dose of 70 Gy/ 25 fractions of a single daily dose of 2.8 Gy. By the linear-quadratic formula, considering an α/β ratio of 1.5 Gy for prostate cancer, 70 Gy/25 fractions is equivalent to 86 Gy in 43 fractions of 2 Gy. All patients were simulated on CT simulator.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — The IMRT plan consisted of five - seven fields to deliver the same dose prescribed at the isodose line covering 95% of PTV.
  The 3DCRT plan consisted of six fields to deliver a total dose of 70 Gy/ 25 fractions of a single daily dose of 2.8 Gy.
  Other Names: 3DCRT

SUMMARY:
There is no randomized controlled trial (RCT) comparing Conformal Radiotherapy (3DCRT) versus the Intensity Modulated Radiotherapy (IMRT) in terms of toxicity and disease control. Data from retrospective studies show that IMRT reduces the risk of severe late complications. More recently, the results from the RTOG 0126 study have also confirmed the benefit from IMRT in reducing acute toxicity for prostate cancer treated with conventional dose escalation. Therefore, to investigate the real clinical benefit of the IMRT over 3DCRT using a hypofractionated schedule in prostate cancer, the investigators developed a RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of prostate cancer
* With age between 18-75 years classified in low
* Intermediate and high-risk group according to their Gleason score
* T stage and initial PSA (iPSA).
* Low risk group included patients with Gleason score <7 / stage T1-T2a, and iPSA <10 ng/mL.
* Intermediate risk included Gleason score < 7, or Stage T1-T2b, or iPSA level of 10-20 ng/mL
* High-risk patients with Gleason score >7, or Stage > T2b, or iPSA >20 ng/mL.
* All patients classified as high risk was submitted to the bone scans.

Exclusion Criteria:

* Patients with metastases
* Prior history of prostatectomy
* Pelvic radiotherapy treatment
* Chemotherapy treatment were excluded of this trial.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal and geniturinary acute toxicity | 6 months
  The primary study outcome was acute treatment reactions from the beginning of treatment to 6 months after the end of treatment. Patients were seen weekly, or as required, during treatment by a radiation oncologist. Acute gastrointestinal (GI) and genitourinary (GU) toxicity were prospectively assessed and graded according to the Radiation Therapy Oncology Group scoring system for the rectum and bladder.
Gastrointestinal and geniturinary late toxicity | 24 months
  Any toxicity developed after 6 months from radiotherapy treatment was considered as late toxicity. Late gastrointestinal (GI) and genitourinary (GU) toxicity were prospectively assessed and graded according to the Radiation Therapy Oncology Group scoring system for the rectum and bladder.

SECONDARY OUTCOMES:
Biochemical control | 3 years
  The Phoenix criteria ( nadir + 2 ng/ml of PSA) was used to define the biochemical control.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Viani, PhD, Principal Investigator — FAMEMA
Locations (1):
- Faculty of Medicine of Marilia, Marília, São Paulo, Brazil